CLINICAL TRIAL: NCT03701217
Title: Eltrombopag Used in Thrombocytopenia After Comsolidation Therapy in Acute Myeloid Leukemia (AML)
Brief Title: Eltrombopag Used in Thrombocytopenia After Comsolidation Therapy in AML
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Second Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Southern Medical University, China (Other); Wuhan General Hospital of Guangzhou Military Command (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Dongguan Kanghua Hospital (Other)
Responsible Party: Principal Investigator, Dan Xu, professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Eltrombopag-AML-2018
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Eltrombopag; Thrombocytopenia; Acute Myeloid Leukemia
MeSH Terms: conditions — Thrombocytopenia; Leukemia, Myeloid, Acute | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eltrombopag treatment (Experimental): Eltrombopag 25mg bid, starts from the day when platelet count decreases lower than 30×10'9/L, and the treatment lasts for at least 5 days, and stops until platelet count goes up to more than 30×10'9/L, after consolidation therapy in AML patents. Platelet transfusion application is routinely done when platelet count is lower than 20×10'9/L or active hemorrage happens to patients.
  Interventions: Drug: Eltrombopag
- Eltrombopag free (Active Comparator): Eltrombopag treatment is not performed in this group. Platelet transfusion application is routinely done when platelet count is lower than 20×10'9/L or active hemorrage happens to patients.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag 25mg bid, starts from the day when platelet count decreases lower than 30×10'9/L, and the treatment lasts for at least 5 days, and stops until platelet count goes up to more than 30×10'9/L, after consolidation therapy in AML patents.

SUMMARY:
Eltrombopag has been used in the treatment of immune thrombocytopenia (ITP), and significantly increased platelet count and decreased fatal hemorrage. As it's known that all patients with acute leukemia will experience bone marrow suppression and thrombocytopenia after chemotherapy. Some patients even died of fatal bleeding during this period for lacking of platelet transfusion or platelet transfusion refractoriness. So a lot needs to be done to shortern thrombocytopenia time or reduce fatal hemorrage incidence after chemotherapy in acute leukemia patients. In this prospective randomized controlled study, the effect and safety of eltrombopag in the treatment of thrombocytopenia after consolidation therapy in acute myeloid leukemia (AML) is evaluated.

DETAILED DESCRIPTION:
Eltrombopag has been used in the treatment of immune thrombocytopenia (ITP), and significantly increased platelet count and decreased fatal hemorrage. As it's known that all patients with acute leukemia will experience bone marrow suppression and thrombocytopenia after chemotherapy. Some patients even died of fatal bleeding during this period for lacking of platelet transfusion or platelet transfusion refractoriness. So a lot needs to be done to shortern thrombocytopenia time or reduce fatal hemorrage incidence after chemotherapy in acute leukemia patients. In this prospective randomized controlled study, the effect and safety of eltrombopag in the treatment of thrombocytopenia after consolidation therapy in acute myeloid leukemia (AML) is evaluated.

ELIGIBILITY:
Inclusion Criteria:

All patients with the age range from 14 to 60 years old with AML exclusive of APL in CR status; All those accepting IA or DA (IDA 10mg or DNR 45mg/m2, d1-3, Ara-C 2g/m2 q12h, d1-3) or MDAC (Ara-C 2g/m2 q12h, d1-3) as consolidation regimens.

Exclusion Criteria:

Those without obtaining CR; Those experience more 6 cycles of chemotherapy; Any abnormality in a vital sign (e.g., organ function failure, serious infection ); Patients with any conditions not suitable for the trial (investigators' decision).

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Thrombocytopenia time | 30 days after consolidation therapy.
  The lasting time for platelet count lower than 20×10'9/L after consolidation therapy.
The incidence of fatal hemorrage | 30 days after consolidation therapy.
  Fatal hemorrage includes all bleedings have life-threaten to the patients, eg. gastrointestinal bleeding, brain bleeding, pneumorrhagia, etc.

SECONDARY OUTCOMES:
The incidence of thrombus | 30 days after consolidation therapy.
  All kinds of thrombus happens in veins and arteries after consolidation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Xu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided